CLINICAL TRIAL: NCT04515342
Title: Sarcopenia, Fall and Osteoporosis in Patients With Chronic Kidney Disease
Brief Title: Sarcopenia, Fall and Osteoporosis in Chronic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Ditte Hansen, Associate professor, MD, PhD, Herlev Hospital
Other Study IDs: SarcoCKD2020
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Sarcopenia; Chronic Kidney Diseases; Osteoporosis
Keywords: Fall; Chronic kidney disease-mineral and bone disorder (CKD-MBD)
MeSH Terms: conditions — Sarcopenia; Renal Insufficiency, Chronic; Osteoporosis; Bone Diseases; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Muscle Strength; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples (serum, plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: This is a cross-sectional study involving approximately 150 patients. They undergo a physical examination, fill out a questionnaire, have blood samples drawn, undergo a Dual Energy X-ray Absorptiometry (DXA) scan and different physical procedures to assess muscle strength and muscle function.
  Interventions: Diagnostic Test: DXA; Other: Muscle strength and function assessment; Other: Blood samples

INTERVENTIONS:
Diagnostic Test: DXA — Each participant will undergo one DXA scan
Other: Muscle strength and function assessment — Each patient will have their muscle strength and function assessed with the measurements of handgrip strength, 10 m gait speed and a 30 s sit-to-stand test. They will also fill out a questionnaire assessing Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls (SARC-F questionnaire).
Other: Blood samples — Each patient will undergo a physical examination and also deliver blood samples.

SUMMARY:
This study is a cross-sectional study that wishes to investigate whether there is an increased incidence of sarcopenia in patients with chronic kidney disease compared to the Danish background population. A possible association between sarcopenia and fall, as well as the incidence of osteoporosis in patients with chronic kidney disease will also be described.

DETAILED DESCRIPTION:
Sarcopenia is a condition diagnosed from different clinical findings such as low muscle mass, low muscle strength and possibly also poor physical performance. In the general population, the risk of fall and bone fracture increases, when sarcopenia is also present.

Sarcopenia is known to occur in patients with chronic kidney disease, but whether, and if so, how this differs from the incidence in patients without kidney disease has not previously been described.

Patients with chronic kidney disease have a 3 times higher risk of bone fracture compared to the Danish background population, and they also have an increased risk of falls.

The association between sarcopenia, risk of falls and osteoporosis in patients with kidney disease is until now sparsely described, and because of this, the investigators want to explore this further in this cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Chronic kidney disease stage 4-5 not on dialysis (nonD) (corresponding to an estimated glomerular filtration rate (eGFR) ≤30 ml/min based on Kidney Disease Improving Global Outcomes (KDIGO) definition and not on dialysis)

Exclusion Criteria:

* Kidney transplanted
* Immobilized/hospitalized for more than 1 week within the last 6 weeks
* Active treatment with growth hormone or sex hormone
* Known muscle disease
* The lack of ability to speak or understand Danish
* The lack of ability to give an informed consent
* The lack of ability to participate in a clinical study based on the assessment by the local investigator

Ages: 20 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the Department of Nephrology at both Herlev Hospital and Odense University Hospital during their regular visits to these outpatient clinics.
  All subjects connected to the participating centers are screened to see if they are eligible for the study. Participants with a minimum age of 20 with eGFR ≤30 ml/min are asked if they wish to be examined further to see if they meet all the inclusion criteria and none of the exclusion criteria. Only participants meeting all the inclusion criteria and none of the exclusion criteria will be considered eligible for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference in appendicular lean body mass | Day 0 (day of study procedure)
  Difference in appendicular lean body mass between patients with chronic kidney disease and a healthy control group examined in a previous study

SECONDARY OUTCOMES:
Difference in the incidence of sarcopenia | Day 0 (day of study procedure)
  Difference in the incidence of sarcopenia between patients with chronic kidney disease and a healthy control group examined in a previous study
Difference in appendicular muscle mass | Day 0 (day of study procedure)
  Difference in appendicular muscle mass between patients with chronic kidney disease and a healthy control group examined in a previous study
Difference in handgrip strength | Day 0 (day of study procedure)
  Difference in handgrip strength between patients with chronic kidney disease and a healthy control group examined in a previous study
Difference in gait speed | Day 0 (day of study procedure)
  Difference in gait speed between patients with chronic kidney disease and a healthy control group examined in a previous study
Difference in sit-to-stand test | Day 0 (day of study procedure)
  Difference in sit-to-stand test between patients with chronic kidney disease and a healthy control group examined in a previous study
Difference in the incidence of osteoporosis | Day 0 (day of study procedure)
  Difference in the incidence of osteoporoses between patients with chronic kidney disease and a healthy control group examined in a previous study
Difference in the tendency to fall | Day 0 (day of study procedure)
  Difference in the tendency to fall between patients with chronic kidney disease and a healthy control group examined in a previous study
The correlation between total lean and appendicular lean body mass, handgrip strength, gait speed, sit-to-stand test, tendency to fall and osteoporosis | Day 0 (day of study procedure)
  The correlation between total lean and appendicular lean body mass, handgrip strength, gait speed, sit-to-stand test, tendency to fall and osteoporosis (T-score <-2.5 in hip and/or lumbal spine)

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, MD, PhD, Principal Investigator — Department of Nephrology, Herlev and Gentofte Hospital
Locations (2):
- Denmark (2):
  - Herlev and Gentofte Hospital, Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
For now no Individual Participant Data (IPD) are planned to be shared with other researchers.

REFERENCES:
- [Background] Suetta C, Haddock B, Alcazar J, Noerst T, Hansen OM, Ludvig H, Kamper RS, Schnohr P, Prescott E, Andersen LL, Frandsen U, Aagaard P, Bulow J, Hovind P, Simonsen L. The Copenhagen Sarcopenia Study: lean mass, strength, power, and physical function in a Danish cohort aged 20-93 years. J Cachexia Sarcopenia Muscle. 2019 Dec;10(6):1316-1329. doi: 10.1002/jcsm.12477. Epub 2019 Aug 16. PMID 31419087